CLINICAL TRIAL: NCT03844503
Title: Food Prototype Containing Resistant Starch Type 4 on Postprandial Glycemic Response in Healthy Adults
Brief Title: Food Containing Resistant Starch Type 4 and Postprandial Glycemic Response
Acronym: RS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB2019-005
Record Dates: First submitted 2019-02-05; First posted 2019-02-18 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Cereal bar; Fiber; Resistant Starch; Glycemic Response; Insulin Response
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cereal Bar no fiber (Placebo Comparator): Cereal bar without fiber
  Interventions: Dietary Supplement: Cereal Bar no fiber
- Cereal bar with 10 g fiber (Active Comparator): Cereal bar with 10 g fiber
  Interventions: Dietary Supplement: Cereal bar with 10 g fiber
- Cereal bar with 20 g fiber (Active Comparator): Cereal bar with 20 g fiber
  Interventions: Dietary Supplement: Cereal bar with 20 g fiber

INTERVENTIONS:
Dietary Supplement: Cereal Bar no fiber — Cereal Bar no fiber
  Arms: Cereal Bar no fiber
Dietary Supplement: Cereal bar with 10 g fiber — Cereal bar with 10 g fiber
  Arms: Cereal bar with 10 g fiber
Dietary Supplement: Cereal bar with 20 g fiber — Cereal bar with 20 g fiber
  Arms: Cereal bar with 20 g fiber

SUMMARY:
The primary objective of the study is to determine if resistant starch reduces the 2 hour glycemic response as measured by positive incremental area under the blood glucose response curve (Positive iAUC- ignores area below fasting). Secondary endpoints include insulin iAUC, glucose and insulin net incremental AUC (net iAUC), time point of peak rise (T max) of glucose and insulin, and glucose and insulin concentrations at each time point (C max).

DETAILED DESCRIPTION:
This is a single-center randomized, single-blinded, cross-over design study to allow for three acute evaluations of 2 hr postprandial glucose in response to 3 cereal bars containing different amounts of resistant starch. The study will evaluate acute glucose and insulin response in healthy men and women aged 20-45 years.

The trial will initiate with record collection to assess background general health (screening visit) and dietary intake followed by counseling to follow a relatively low polyphenolic beverages/foods diet, and high fiber containing food (particularly fermentable) which will commence at least 3 days before randomization (washout) and continue for the duration of the study. After 3-day washout period, subjects will be randomized to treatment order within Phase (Treatment cereal bars A, B, C). Glucose and insulin responses following the consumption of cereal bars will be determined by blood collections via venous catheter. Blood samples (3 ml of blood) will be collected at -5 min (before the cereal bar consumption) and 15, 30, 45, 60, 90, and 120 min after consuming bars for assessment in changes in glucose and insulin concentrations in the plasma. The primary endpoint is glucose positive incremental area under the curve (positive iAUC- ignores area below fasting) among the three tests bars. Secondary endpoints are glucose peak, insulin positive iAUC and peak and glucose and insulin net incremental AUC (net iAUC). Adverse events also will be collected and frequency tabulated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female, 20-45 years of age, inclusive.
* Subject has a BMI of 20.0-24.9 kg/m2, inclusive and weight ≥ 110 lb. at screening visit.
* Subject is willing to maintain his/her usual physical activity pattern throughout the study period.
* Subject is willing to follow study instructions including compliance with dietary restrictions, consumption of study bars, and study visit schedule.
* Subject is judged to be in good health on the basis of the medical history.
* Subject is willing to abstain from alcohol consumption for 24 hours prior to study visit.
* Exercise to be maintained throughout study duration, including 3 days before study visit
* Subject is willing to maintain a stable dose of current vitamins, minerals, supplements and medications not interfering with study outcomes, including birth control, throughout the study duration.
* Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator/s and is willing to complete study procedures.

Exclusion Criteria:

* Subject has fasting finger prick glucose >100 mg/dL.
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at the screening visit.
* Subject has had major trauma or a surgical event within 2 months of study visit 1.
* Subject has had a weight change ≥4.5 kg within 2 months of visit, taking weight loss drugs, or has had bariatric surgery or other weight reduction surgery (i.e. liposuction, laser fat removal, etc)
* Subject has a history or presence of clinically important endocrine, cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary, or gastrointestinal disorders that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
* Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Subject has a history of extreme dietary habits, as judged by the Investigator (e.g., Atkins diet, etc.).
* Subject has a history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
* Subject has a known intolerance or sensitivity to any ingredients in the study products.
* Subject has used medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, hypoglycemic medications, and systemic corticosteroids 2 weeks prior to visit 1 and throughout the study.
* Subjects who used fiber supplements.
* Subject taking systemic steroids, extreme alcohol use, or drug user.
* Subject has vein access score less than 7.
* Subject is a female, who is pregnant, planning to be pregnant during the study period or lactating.
* Subject is a current smoker. Past smoker abstinence for less than 2 years.
* Subject has participated in any clinical trial within 30 days prior to enrollment.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Changes in Plasma Glucose concentration as measured by positive incremental area under the curve (positive iAUC) over 2 hours | Postprandial 2 hours
  Changes in plasma glucose concentration as measured by positive iAUC (ignoring area below fasting) over a 2 hour Postprandial Test day after administration of active treatment compared to control treatment

SECONDARY OUTCOMES:
Changes in plasma insulin concentration as measured by iAUC over a 2 hour Postprandial Test day after administration of active treatments compared to control treatment | Postprandial 2 hours
  Changes in plasma insulin concentration as measured by iAUC over a 2 hour Postprandial Test day after administration of active treatment compared to control treatment
Changes in Plasma Insulin concentration as measured by positive incremental area under the curve (positive iAUC) over 2 hours | Postprandial 2 hours
  Changes in Plasma Insulin concentration as measured by positive incremental area under the curve (positive iAUC) over 2 hours
Plasma Glucose maximal concentration (Cmax) over 2 hours | Postprandial 2 hours
  Plasma Glucose maximal concentration (Cmax) over 2 hours
Plasma Insulin maximal concentration (Cmax) over 2 hours | Postprandial 2 hours
  Plasma Insulin maximal concentration (Cmax) over 2 hours
Change in postprandial blood glucose concentration responses for treatments compared to control over 2-hour postprandial period | Postprandial 2 hours
  postprandial blood glucose concentration responses over 2 hours
Change in postprandial blood insulin concentration responses for treatments compared to control over 2-hour postprandial period | Postprandial 2 hours
  postprandial blood insulin concentration responses over 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided